CLINICAL TRIAL: NCT04219878
Title: Engaging African American and Hispanic/Latino MSM for HIV Testing and Prevention Services Through Technology
Brief Title: Implementation of Rapid HIV Self-Testing Among MSM Project
Acronym: iSTAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Patrick S Sullivan, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00099710; 1U01PS005181 (NIH)
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: HIV/AIDS
Keywords: Sexually transmitted infections; Behavioral intervention; Public health; HIV preexposure prophylaxis (PrEP)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Know@Home App or Website and Test Kit (Active Comparator): Participants in this study arm will have access to Know@Home, a mobile HIV prevention app or website and will receive mail-out HIV self-testing kits.
  Interventions: Behavioral: Know@Home; Other: Self-test Kit
- Mail-Out Testing Kit Only (Active Comparator): Participants in this study arm will receive mail-out HIV self-testing kits.
  Interventions: Other: Self-test Kit

INTERVENTIONS:
Behavioral: Know@Home — Participants randomly assigned to the Know@Home arm will access the features of Know@Home by downloading the app or accessing the website. The contents were developed to serve as a comprehensive mobile HIV prevention platform for MSM or TGW, with HIV prevention and care information and links to resources. This intervention arm provides an toolkit that allows users to access information about prevention services as their needs change. Participants will have access to Know@Home for the study period. The Know@Home arm will offer participants the opportunity to order free condoms and lubricant as well as an at-home sexually transmitted infection (STI) testing kit.
  Arms: Know@Home App or Website and Test Kit
Other: Self-test Kit — All participants will be shipped two at-home HIV self-tests. They will also receive a link to a previously-produced video that fully describes the specimen collection process, pointing out common errors and providing tips for successful collection. Participants will interact with study staff through phone, email, or text. Information to schedule a video HIV testing and counseling session with study staff will be made available to participants in all arms via a website, email, and/or text.
  Other Names: OraQuick® In-Home HIV Test

SUMMARY:
This study will use online materials and strategies to recruit 3600 Black and Hispanic men who have sex with men (MSM) and transgender women (TGW) to participate in a study evaluating the effectiveness of the Know@Home mobile app compared to control condition with respect to linkage of participants to appropriate services, as well as cost-effectiveness outcomes.

DETAILED DESCRIPTION:
To evaluate the effectiveness of mailing out rapid HIV home-testing kits and additional testing promotion components among African-American or black and Hispanic or Latino gay, bisexual, and other men who have sex with men (MSM) and transgender women (TGW), the study "Implementation of Rapid HIV Self-Testing among MSM Project", known as iSTAMP, is being conducted in 11 US states. This study is interested in the most cost-effective ways to recruit people at high risk for HIV infection. The researchers want to study a sample of 3600 adult MSM and TGW who are not known to be living with HIV; 1800 black/African-American and 1800 Hispanic/Latino participants will be enrolled.

All participants will be mailed two rapid HIV self-test kits upon randomization. All participants, regardless of study arm, will also complete a follow-up survey at the end of a 4-month follow-up period. At the end of the 4-month follow-up period, participants will be mailed a dried blood spot (DBS) collection kit for research purposes, as well as another rapid HIV self-test kit for immediate testing. Participants in each of the arms will have access to videoconferencing-delivered prevention counseling, and all participants, regardless of assigned arm, will be contacted if they report seroconversion and/or a preliminary positive test during the study period for active linkage to care.

ELIGIBILITY:
Inclusion Criteria for MSM Participants:

* Black/African-American race or Hispanic/Latino ethnicity
* Male sex at birth
* Currently identify as male
* Reported anal sex with at least one man in the past 12 months
* Aged 18 or over
* Has an Android or Apple mobile phone with currently active service
* Currently resides in a study state: North Carolina, South Carolina, Georgia, Alabama, Mississippi, Florida, Louisiana, California, Nevada, Texas, New York
* Willing to download a study participation management mobile app
* Willing to provide valid contact information so that study HIV testing kits and other materials (condoms, lubricants, STI testing kits) can be mailed to participants.
* Successful completion of baseline survey

Exclusion Criteria for MSM Participants:

* Currently participating in another HIV prevention research study or program
* Has a bleeding disorder preventing use of dried blood spot testing
* Has previously participated in an HIV vaccine study.
* Currently taking PrEP for HIV prevention
* Self-reports living with HIV
* Has plans to move out of a study state during the study period (4 months)

Inclusion Criteria for TGW:

* Male sex at birth
* Currently identify as transgender woman or female
* Aged 18 or over
* Has an Android or Apple mobile smartphone with currently active service
* Currently resides in a study state: North Carolina, South Carolina, Georgia, Alabama, Mississippi, Florida, Louisiana, California, Nevada, Texas, New York
* Willing to provide valid contact information so that study HIV testing kits and other materials (condoms, lubricants, STI testing kits) can be mailed to participants
* Successful completion of baseline survey

Exclusion Criteria for TGW:

* Currently participating in another HIV prevention clinical trial or intervention
* Has a bleeding disorder preventing use of dried blood spot testing
* Has previously participated in an HIV vaccine study
* Currently taking PrEP for HIV prevention
* Self-reports living with HIV
* Has plans to move out of a study state during the study period (4 months)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study includes participants who were assigned male sex at birth and identify as male or female.
Enrollment: 2195 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Number of participants initiating HIV treatment | Up to Month 4
  Effectiveness of the interventions will be assessed by linkage of participants to HIV treatment.
Number of participants initiating PrEP treatment | Up to Month 4
  Effectiveness of the interventions will be assessed by linkage of participants to PrEP treatment.
Number of participants testing for STIs | Up to Month 4
  Effectiveness of the interventions will be assessed by linkage of participants to STI testing.
Number of participants engaging in HIV prevention services | Up to Month 4
  Effectiveness of the interventions will be assessed by linkage of participants to HIV prevention services.
Number of participants engaging in HIV social services | Up to Month 4
  Effectiveness of the interventions will be assessed by linkage of participants to HIV social services.
Cost of different online venues for study enrollment | Baseline
  Enrollment in the study defined as completion of the baseline survey and downloading of the study app. The cost (in US dollars) to enroll participants (online banner advertisement placement, study staff time to manage enrollment, validating participant eligibility, monitoring and evaluation of enrollment data) will be compared between the study arms.
Cost of different online venues for HIV test results returned | Month 1
  The cost (in US dollars) of HIV tests returned within 1 month of enrollment will be compared between the study arms. The costs involved with having HIV tests returned include:
  * Online banner advertisement placement
  * Study staff time managing enrollment, validating participant eligibility, monitoring and evaluation of enrollment data
  * HIV test kits
  * Shipping for HIV test kits
  * Staff/personnel time to manage mailing/return of test kits
  * Other general and administrative time, office supplies, equipment, rents, utilities
Cost of different online venues for identifying new HIV diagnoses | Month 1
  The cost (in US dollars) of identifying established HIV infections will be compared between the study arms. The costs involved with identifying established HIV infections include:
  * Online banner advertisement placement
  * Study staff time managing enrollment, validating participant eligibility, monitoring and evaluation of enrollment data
  * HIV test kits
  * Shipping for HIV test kits
  * Staff/personnel time to manage mailing/return of test kits
  * Study staff time to manage monitoring and evaluation of HIV test result data
  * Study staff time to provide phone counseling to those with established infections
  * Other general and administrative time, office supplies, equipment, rents, utilities

SECONDARY OUTCOMES:
Cost of linkage to HIV counseling | Month 4
  The cost (in US dollars) of linking participants testing positive for HIV to HIV counseling will be compared between the study arms, including:
  * Study staff time spent contacting participants
  * Study staff time for intervention maintenance (e.g., app management)
  * HIV counseling costs to the healthcare system
  * Other general and administrative time, office supplies, equipment, rents, utilities
Cost of linkage to HIV treatment | Month 4
  The cost (in US dollars) of linking participants testing positive for HIV to HIV treatment will be compared between the three study arms, including:
  * Study staff time for intervention maintenance (e.g., app management)
  * HIV treatment costs to the healthcare system
  * Other general and administrative time, office supplies, equipment, rents, utilities
Cost of linkage to PrEP counseling | Month 4
  The cost (in US dollars) of linking participants testing negative for HIV to PrEP counseling will be compared between the study arms, including:
  * Study staff time contacting participants
  * Study staff time for intervention maintenance (e.g., app management)
  * PrEP counseling costs to the healthcare system
  * Other general and administrative time, office supplies, equipment, rents, utilities
Cost of linkage to PrEP uptake | Month 4
  The cost (in US dollars) of linking participants testing negative for HIV to initiate PrEP treatment will be compared between the study arms, including:
  * Study staff time contacting participants
  * Study staff time for intervention maintenance (e.g., app management)
  * PrEP uptake costs to the healthcare system
  * Other general and administrative time, office supplies, equipment, rents, utilities
Cost of Sexually Transmitted Infection (STI) testing | Month 4
  The cost (in US dollars) of providing at-home STI testing be compared between the study arms, including:
  * Cost of STI testing materials and shipping
  * Laboratory STI testing
  * Study staff time processing orders and contacting participants
  * Study staff time for intervention maintenance (e.g., app management)
  * STI testing costs to the healthcare system
  * Other general and administrative time, office supplies, equipment, rents, utilities
Cost of linkage to STI treatment | Month 4
  The cost (in US dollars) of providing treatment for STIs discovered through at-home STI testing be compared between the three study arms, including:
  * Study staff time processing orders and contacting participants
  * Study staff time for intervention maintenance (e.g., app management)
  * STI treatment costs to the healthcare system
  * Other general and administrative time, office supplies, equipment, rents, utilities

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Sullivan, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial will be available for sharing with other researchers, after deidentification. Some data may be provided as categorical variables.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available 30 months after data collection and cleaning have ended until five years after data are made available.
Access Criteria: Data will be available to anyone affiliated with public health organizations, agencies or accredited universities requesting to access the data for any research purpose that is approved by the Centers for Disease Control and Prevention (CDC) Project Officer and Emory University Principal Investigator. Proposals should be directed to rmacgowan@cdc.gov. To gain access, data requestors must work as a member of the study team on data analysis and manuscript preparation.

REFERENCES:
- [Derived] MacGowan RJ, Chavez PR, Dana R, Hannah M, Raiford JL, Caldwell JA, Wall KM, Johnson JA, Sharma A, Hightow-Weidman L, Stephenson R, Sanchez T, Smith AJ, Sullivan S, Jones J, Sullivan PS. Efficacy of Internet Recruitment and HIV Self-Testing for Diagnosing HIV Infections Among Black and Hispanic/Latino MSM and Transgender Women in 11 US States, 2020-2021. J Acquir Immune Defic Syndr. 2024 Oct 1;97(2):133-141. doi: 10.1097/QAI.0000000000003476. PMID 39250647
- [Derived] Dana R, Sullivan S, MacGowan RJ, Chavez PR, Wall KM, Sanchez TH, Stephenson R, Hightow-Weidman L, Johnson JA, Smith A, Sharma A, Jones J, Hannah M, Trigg M, Luo W, Caldwell J, Sullivan PS. Engaging Black or African American and Hispanic or Latino Men Who Have Sex With Men for HIV Testing and Prevention Services Through Technology: Protocol for the iSTAMP Comparative Effectiveness Trial. JMIR Res Protoc. 2023 Jan 6;12:e43414. doi: 10.2196/43414. PMID 36607707

DOCUMENTS (1):
  • Informed Consent Form (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT04219878/ICF_000.pdf